CLINICAL TRIAL: NCT02535780
Title: Novel Transcranial Treatments to Modulate Taste Reward and Body Perception Pathways in Eating Disorders
Brief Title: Transcranial Treatments in Eating Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study procedures and time not feasible due to patient schedule
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2716
Record Dates: First submitted 2015-08-06; First posted 2015-08-31 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- TMS Treatment Group (Experimental): 15 sessions active Transcranial magnetic stimulation (TMS) treatment
  Interventions: Procedure: Transcranial magnetic stimulation
- TMS Sham Group (Sham Comparator): 15 sessions sham Transcranial magnetic stimulation (TMS) treatment
  Interventions: Procedure: Transcranial magnetic stimulation
- tDCS Treatment Group (Experimental): 15 sessions active Transcranial direct current stimulation (tDCS) treatment
  Interventions: Procedure: Transcranial direct current stimulation
- tDCS Sham Group (Sham Comparator): 15 sessions sham Transcranial direct current stimulation (tDCS) treatment
  Interventions: Procedure: Transcranial direct current stimulation

INTERVENTIONS:
Procedure: Transcranial magnetic stimulation — TMS
  Arms: TMS Sham Group; TMS Treatment Group
Procedure: Transcranial direct current stimulation — tDCS
  Arms: tDCS Sham Group; tDCS Treatment Group

SUMMARY:
The primary aim of this study is to study how Repetitive Transcranial Magnetic Stimulation (rTMS) tailored to specific anorexia nervosa (AN) or bulimia nervosa (BN) brain activation alterations will promote recovery and to study how inhibitory tDCS (Transcranial Direct Current Stimulation) will reduce symptoms of body image distortion in a second sample of AN and BN groups.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa subjects:
* Meets DSM-5 criteria for anorexia nervosa (AN) either binge-eating/purging type or restricting-type:
* Intense fear of gaining weight or becoming fat, even though underweight.
* The ability to undergo an MRI, fMRI or other similar procedure requiring spending time in an enclosed space
* Bulimia Nervosa subjects:
* Meet DSM-5 criteria for bulimia nervosa (BN):
* Self-induced vomiting; misuse of laxatives, diuretics, enemas, medication, fasting, excessive exercise.

Exclusion Criteria:

* Electrolyte, blood count or kidney or liver function abnormalities.
* No symptoms of alcohol or other substance abuse or dependence in the past 3 months,
* No previous or current organic brain syndromes, dementia, psychotic disorders, somatization disorders, or conversion disorder, head trauma, indication of mental retardation or pervasive developmental disorder.
* No antipsychotics, tricyclic antidepressants or Wellbutrin or other medication that may lower the seizure threshold.
* Claustrophobia.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
taste reward brain function activation confirmed by Functional magnetic resonance imaging (fMRI) | 3 years
  Change in brain activation to taste reward paradigm

SECONDARY OUTCOMES:
Change in self-reported measures related to eating disorder thoughts and behaviors | 3 years
  Self Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Guido K. Frank, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver and Health Science Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No